CLINICAL TRIAL: NCT02484508
Title: A Randomized, Double Blind, Single Simulation, Parallel Controlled, Multi-center Clinical Study of Guli Capsules in the Treatment of Knee Osteoarthritis
Brief Title: Multi-center Clinical Study of Guli Capsules in the Treatment of Knee Osteoarthritis
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Guizhou Bailing Group Pharmaceutical Co Ltd (Industry)
Collaborators: Wangjing Hospital, China Academy of Chinese Medical Sciences (Other); The First Affiliated Hospital of Guiyang College of Traditional Chinese Medicine (Unknown); People's Hospital of Anshun City of Guizhou Province (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: GL-15-01
Record Dates: First submitted 2015-06-16; First posted 2015-06-29 (Estimated); Last update posted 2015-06-29 (Estimated); Status verified 2015-06

CONDITIONS: Knee Osteoarthritis
Keywords: Guli capsule; knee osteoarthritis; Changing of WOMAC and VAS score
MeSH Terms: conditions — Osteoarthritis, Knee

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Guli capsule (Experimental): Guli capsule, the tested drug of this study
  Interventions: Drug: Guli capsule
- Kangguzengsheng capsule (Active Comparator): Kangguzengsheng capsule, a CFDA approved drug for articular genu osteoarthritis,is adopted as active comparator in this study
  Interventions: Drug: Kangguzengsheng capsule

INTERVENTIONS:
Drug: Guli capsule — Guli capsule,as the experimental drug,is taken 3 grains each time, 3 time per day
  Other Names: GL capsule
  Arms: Guli capsule
Drug: Kangguzengsheng capsule — Kangguzengsheng capsule, as the active comparator, is taken 3 grains each time, 3 time per day
  Other Names: KGZS capsule
  Arms: Kangguzengsheng capsule

SUMMARY:
Previous study showed that Guli capsule could suppress the adjuvant multiple arthritis; have inhibitory effect on carrageenan gelatinous and formaldehyde foot swelling; improve the symptom of osteoporosis patients; and improve pain and limited joint activities of rheumatoid patients.

To further verify the clinical effect of Guli capsule in the treatment of knee osteoarthritis, the investigators perform this multi-center clinical study.

DETAILED DESCRIPTION:
Guli capsule, an approved Chinese patent drug, its main indications are for rheumatism, rheumatoid arthritis.

Previous study showed that Guli capsule could suppress the adjuvant multiple arthritis; have inhibitory effect on carrageenan gelatinous and formaldehyde foot swelling; improve the symptom of osteoporosis patients; and improve pain and limited joint activities of rheumatoid patients.

To further verify the clinical effect of Guli capsule in the treatment of knee osteoarthritis, the investigators perform this multi-center clinical study.

ELIGIBILITY:
Inclusion Criteria:

* Ages between 40 and 70 years, both gender
* Kellgren and Lawrence grades of I to III;
* The subjects volunteered participate in the study and complied with the regulations and signed the written consent voluntarily.
* Meet the following clinical and radiological criteria for diagnosis:
* Clinical criteria:

  1. most of the time have knee pain nearly a month
  2. bone fricative
  3. morning stiffness is less than or equal to 30 min
  4. age is more than or equal to 38 years
  5. bony enlargement. Who meet (1) + (2) or (1) + (4) + (5) can be diagnosed as knee osteoarthritis.
* Radiological criteria:

  1. most of the time have knee pain nearly a month
  2. the X-ray showed osteophyte formation
  3. joint fluid examination confirmed with osteoarthritis
  4. age is more than or equal to 40 years
  5. morning stiffness is less than or equal to 30 min
  6. bone fricative. Meet (1) + (2) or (1) + (3) + (5) + (6) or (1) + (4) + (5) + (6).

Exclusion Criteria:

* Patient with a history of allergy to similar constituents or chemical components of the drug;
* Patients with limited liver and kidney function;
* Patients with hematopoietic system disease;
* Patients with diabetes, Cushing's syndrome and other endocrine disorders;
* Patients with severe heart and brain disease;
* Patients with low immunity;
* Patients directly involved with the staff in the study;
* Women during pregnancy or lactation;
* Participating in other clinical studies or Participated in 3 months;
* The investigators judged who be unfit for the study.

Ages: 40 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 220 (Estimated)
Dates: Start 2015-03; Primary Completion 2016-03 (Estimated); Study Completion 2016-03 (Estimated)

PRIMARY OUTCOMES:
Osteoarthritis index on the Western Ontario and McMaster Universities Osteoarthritis Index | 4 weeks

SECONDARY OUTCOMES:
Pain Scores on the Visual Analog Scale | 4 weeks
Number of Participants with Adverse Events as a Measure of Safety | 4 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Weiheng Chen, MD Dr., Principal Investigator — ICMJE
Locations (1):
- Wangjing Hospital, Chinese Academy of Traditional Chinese Medicine, Beijing, Beijing Municipality, China